CLINICAL TRIAL: NCT02707484
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Study of Efficacy of Thalidomide for Refractory Small Intestinal Bleeding From Vascular Malformation
Brief Title: the Efficiency of Thalidomide for Recurrent Small Intestinal Bleeding Due to Gastrointestinal Vascular Malformation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Peking Union Medical College Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Xinqiao Hospital of Chongqing (Other); Changhai Hospital (Other); Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Director of digestive endoscopy center of Renji hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rj(2015)088K-a
Record Dates: First submitted 2015-11-17; First posted 2016-03-14 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Vascular Malformation
Keywords: Gastrointestinal vascular malformation; thalidomide; Small intestinal bleeding
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thalidomide Group（100mg） (Experimental): Generic name:Thalidomide Dosage form:tablet, 25mg Dosage:100mg/day Frequency: 25mg, QID, Oral Duration:120 days
  Interventions: Drug: Thalidomide (100mg)
- Thalidomide Group（50mg） (Experimental): Generic name:Thalidomide Dosage form:tablet, 25mg&Placebo Dosage:50mg/day Frequency: 25mg BID &Placebo, BID, Oral Duration:120 days
  Interventions: Drug: Thalidomide (50mg)
- placebo -controlled Group (Placebo Comparator): Generic name:Thalidomide Placebo Dosage form:tablet, Placebo Dosage:Placebo Frequency: Placebo, QID, Oral Duration:120 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Thalidomide (100mg) — Patients were randomly assigned to receive a 120-days course of 100 mg of thalidomide (Pharmaceutical Co., Ltd. of ChangZhou, China).
  Other Names: Group 1
  Arms: Thalidomide Group（100mg）
Drug: Thalidomide (50mg) — Patients were randomly assigned to receive a 120-days course of 50 mg of thalidomide (Pharmaceutical Co., Ltd. of ChangZhou, China).
  Other Names: Group 2
  Arms: Thalidomide Group（50mg）
Drug: placebo — Patients were randomly assigned to receive a 120-days course of placebo (Pharmaceutical Co., Ltd. of ChangZhou, China).
  Other Names: Group 3
  Arms: placebo -controlled Group

SUMMARY:
Gastrointestinal vascular malformation (GIVM), which is an important cause of acute or chronic gastrointestinal bleeding, currently lacks of effective treatment. The investigators' previous study first confirmed thalidomide treatment of GIVM bleeding was safe and effective. This prospective multi-center randomized controlled clinical trial intends to investigate the efficacy of thalidomide to the recurrent small intestinal hemorrhage due to GIVM.

DETAILED DESCRIPTION:
This multi-institutional clinical trial investigates the efficacy of thalidomide to the recurrent small intestinal hemorrhage due to GIVM. Patients with annual average bleeding 4 times or more and lesions located in the small intestine which are not suitable for endoscopic therapy will be randomly assigned to receive A(25mg,Thalidomide，qid), B(25mg, Thalidomide, bid& placebo bid ) or placebo(deferred treatment group) for 4 months. The primary endpoints were the effective response of patients with ≥50% reduction of numbers of bleeding episodes, followed by rate of cases with cessation of bleedin, the difference in blood transfusion, hospitalization, transfusion volume of red cell, average bleeding duration, average hemoglobin level, yearly hospitalization times, average hospital stay and yearly bleeding episodes. This study will be done at 10 centers in China.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed the informed consent after the nature and the specific procedures of the trial has been verbally explained; they have the opportunity to ask questions.
2. Chinese nationality;
3. Female or male subjects aged 18-75 years. Female subjects must be menopausal or have undergone sterilization such as tubal ligation and hysterectomy, or have no plan to give birth recently and agree to take contraceptive measures such as contraceptive drugs, intrauterine physical birth control rings or contraception condoms; or men must have undergone sterilization or do not plan to have a child recently and agree to take contraceptive measures such as contraceptive drugs, or contraception condoms. These criteria are set to eliminate the risk of subjects of child bearing potential.
4. The subjects must have been diagnosed, by capsule endoscopy and / or balloon-assisted enteroscopy, with small intestinal vascular malformation lesions which are unsuitable or inaccessible to endoscopic therapy or surgical antrectomy. Subjects with persistent, recurrent bleeding, ≥ 4 episodes of overt or occult bleeding over last year.

Exclusion Criteria:

1. Subjects with esophageal varices from cirrhosis of the liver; those with uncontrolled hypertension or hyperglycemia (or diabetics who are being treated with insulin), or those with severe heart (e.g., uncontrolled angina pectoris and / or myocardial infarction, congestive heart failure, etc.), respiratory failure, or renal failure with creatinine (Cr) or blood urea nitrogen (BUN) > 2 times the upper limit of normal (ULN), pancreatic or hepatic disease with abnormal hepatic function with alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin (TBil) > 2 times ULN 3 months before the enrollment, or those with any other diseases that are not suitable for the study as judged by the Investigator;
2. Subjects with a history of severe peripheral neuropathy or seizures, or a history of thromboembolic disease;
3. Subjects who need to continuously use non-steroidal anti-inflammatory drugs, anticoagulants, antiplatelets, acetylsalicylic acid preparations, or Chinese herbal medicines containing ginkgo and echinacea; or those who need to receive other anti-angiogenic drugs for a long time;
4. Subjects with white blood cell counts persistently <3.5 * 10^9 / L;
5. Subjects with a history of small bowel resection;
6. Subjects known or suspected to be allergic to any component of thalidomide；
7. Subjects with severe gastrointestinal bleeding that is life-threatening and requires immediate surgical treatment;
8. Subjects who have previously received thalidomide for gastrointestinal bleeding 30 days before the enrollment;
9. Alcohol and / or substance abusers with addiction or dependence, or those with poor compliance as judged by a doctor;
10. Subjects who participated in other clinical trial 6 months before enrollment;
11. Subjects without legal capacity or self-awareness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
effective response rate | First 1-year follow-up versus the 1-year Observation Period.
  the proportion of patients with "effective treatment, patients with ≥50% reduction of numbers of bleeding episodes after treatment during the First 1-year follow-up versus the 1-year Observation Period.

SECONDARY OUTCOMES:
overall rate of cases with cessation of bleeding | First 1-year follow-up versus the 1-year Observation Period.
  The overall rate of cases with cessation of bleeding without rebleeding during the First 1-year Follow-up Period.
rate of cases requiring blood transfusion | First 1-year follow-up versus the 1-year Observation Period.
  The rate of cases requiring blood transfusion during the First 1-year follow-up.
rate of cases requiring hospitalizations due to bleeding | First 1-year follow-up versus the 1-year Observation Period.
  The rate of cases requiring hospitalizations due to bleeding during the 1st 1-year follow-up
change in the transfusion volume of red cell | First 1-year follow-up versus the 1-year Observation Period.
  The change in the transfusion volume of red cell during the First 1-year Follow-up Period versus the Observation Period.
change in average bleeding duration | First 1-year follow-up versus the 1-year Observation Period.
  The change in average bleeding duration (days) during the First 1-year Follow-up Period versus the Observation Period.
change in average hemoglobin level | First 1-year follow-up versus the 1-year Observation Period.
  The change in average hemoglobin level (g/L) during the First 1-year Follow-up Period versus the Observation Period.
change in yearly hospitalization times | First 1-year follow-up versus the 1-year Observation Period.
  The change in yearly hospitalization times due to bleeding during the First 1-year Follow-up Period versus the Observation Period.
change in average hospital stay | First 1-year follow-up versus the 1-year Observation Period.
  The change in average hospital stay (days)due to bleeding during the First 1-year Follow-up Period versus the Observation Period.
change in yearly bleeding episodes | First 1-year follow-up versus the 1-year Observation Period.
  The change in yearly bleeding episodes during the First 1-year Follow-up Period versus the Observation Period.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Result] Ge ZZ, Chen HM, Gao YJ, Liu WZ, Xu CH, Tan HH, Chen HY, Wei W, Fang JY, Xiao SD. Efficacy of thalidomide for refractory gastrointestinal bleeding from vascular malformation. Gastroenterology. 2011 Nov;141(5):1629-37.e1-4. doi: 10.1053/j.gastro.2011.07.018. Epub 2011 Jul 22. PMID 21784047
- [Result] Ge ZZ, Chen HY, Gao YJ, Hu YB, Xiao SD. Best candidates for capsule endoscopy for obscure gastrointestinal bleeding. J Gastroenterol Hepatol. 2007 Dec;22(12):2076-80. doi: 10.1111/j.1440-1746.2006.04724.x. PMID 18031363
- [Result] Tan H, Chen H, Xu C, Ge Z, Gao Y, Fang J, Liu W, Xiao S. Role of vascular endothelial growth factor in angiodysplasia: an interventional study with thalidomide. J Gastroenterol Hepatol. 2012 Jun;27(6):1094-101. doi: 10.1111/j.1440-1746.2011.06967.x. PMID 22098296
- [Result] Li XB, Ge ZZ, Dai J, Gao YJ, Liu WZ, Hu YB, Xiao SD. The role of capsule endoscopy combined with double-balloon enteroscopy in diagnosis of small bowel diseases. Chin Med J (Engl). 2007 Jan 5;120(1):30-5. PMID 17254484
- [Result] Tan HH, Ge ZZ, Gao YJ, Chen HM, Fang JY, Chen HY, Liu WZ, Xiao SD. The role of HIF-1, angiopoietin-2, Dll4 and Notch1 in bleeding gastrointestinal vascular malformations and thalidomide-associated actions: a pilot in vivo study. J Dig Dis. 2011 Oct;12(5):349-56. doi: 10.1111/j.1751-2980.2011.00506.x. PMID 21955427
- [Result] Feng Q, Tan HH, Ge ZZ, Gao YJ, Chen HM, Xiao SD. Thalidomide-induced angiopoietin 2, Notch1 and Dll4 downregulation under hypoxic condition in tissues with gastrointestinal vascular malformation and human umbilical vein endothelial cells. J Dig Dis. 2014 Feb;15(2):85-95. doi: 10.1111/1751-2980.12114. PMID 24219762
- [Derived] Chen H, Wu S, Tang M, Zhao R, Zhang Q, Dai Z, Gao Y, Yang S, Li Z, Du Y, Yang A, Zhong L, Lu L, Xu L, Shen X, Liu S, Zhong J, Li X, Lu H, Xiong H, Shen Y, Chen H, Gong S, Xue H, Ge Z. Thalidomide for Recurrent Bleeding Due to Small-Intestinal Angiodysplasia. N Engl J Med. 2023 Nov 2;389(18):1649-1659. doi: 10.1056/NEJMoa2303706. PMID 37913505